CLINICAL TRIAL: NCT05482919
Title: The Adolescent Surgery Experience: A Mixed Methods Analysis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 22-019982
Record Dates: First submitted 2022-07-20; First posted 2022-08-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative; Pain; Pain, Acute; Pain, Chronic; Adolescent Behavior; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Pain; Acute Pain; Chronic Pain; Adolescent Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Baseline Survey — The baseline survey, initial PHQ-9 and GAD-7, could be collected prior to surgery after consent, or on the day of surgery, for participants who are undergoing elective surgery or urgent procedures and did not attend pre-operative clinic. Demographic information such as race and ethnicity, pain medications and pain history and baseline self-reported health information will be collected. It will take about 15 minutes to complete.
Behavioral: Post Operative Surveys — Post operative surveys will be collected at one week, two weeks, one month, then monthly up to 6 months after surgery with total of 7 post-op surveys. Refer to Table 1 for visit windows. The study survey could be collected by phone, REDCap texting or email per the subject's preference. Survey content will also include: daily average and maximum self-reported pain scores on a 0-10 Numeric Rating Scale (NRS) pain scale, average hours of sleep, anxiety and depression screens using the PHQ-9 and GAD-7 questionnaires (Months 1, 3, and 5), pain location and quality, percentage of day spent in pain, satisfaction with recovery using a five-point Likert scale, and type, quantity and timing of any medications used for pain (including opioid alternatives).
Behavioral: Qualitative Interviews — Using sampling to identify adolescents who exhibit higher pain scores or prolonged opioid use compared to peers after completion of the first three surveys (pre-operative, Week 1, Week 2), the study will also select a representative sample of adolescents who are recovering as anticipated. Examples of delayed recovery include a higher proportion of moderate to severe pain scores, dissatisfaction with recovery and prolonged opioid use compared to peers. As a balancing measure, the upper limit of adolescents who are perceived to exhibit delayed recovery that are approached for interviews will be capped at a 3:1 ratio compared to those who are recovering as anticipated, and Investigators will prioritize an equal demographic distribution among the two groups. Interviews will take place over the phone or through a CHOP approved vendor at 1 and 3 months after surgery; audio will be recorded with participant consent.

SUMMARY:
New chronic pain and opioid use are reported as prevalent among adolescents undergoing major surgery; many unanswered questions remain regarding recovery and the anticipated pain trajectory across procedures and the interaction between pain treatment, acute inflammation and new chronic pain. Broadly, the proposed study will characterize the adolescent's postoperative recovery experience, and establish the anticipated pain trajectory across a range of procedures.

DETAILED DESCRIPTION:
The proposed study will characterize the adolescent's postoperative pain and recovery experience. Using a mixed methods design, Investigators will follow a diverse cohort of up to 500 adolescents undergoing surgery at the Children's Hospital of Philadelphia (CHOP) over six months to systematically characterize their recovery trajectory. The primary objective is to characterize development of new chronic pain in the context of longitudinal pain trajectories among adolescents in the first 6 months after surgery and to quantify implications of post-surgical pain and pain treatment. The secondary objectives are to determine factors associated with prolonged opioid use after surgery compared to peers (measured in days to discontinuation) and to characterize factors associated with delayed recovery from surgery compared to peers. A baseline survey, including an anxiety and depression screen using the Patient Health Questionnaire-9 (PHQ-9) and General Anxiety Disorder-7 (GAD-7) surveys will be collected after consent and prior to surgery; subsequent post-operative surveys will be collected at one & two weeks, one month, then monthly up to 6 months with total of 8 surveys. The PHQ-9 and GAD-7 will also be administered on month 1, month 3, and month 5. A subgroup of patients will be invited to complete a qualitative interview one month and three months after surgery (+/- 14 days). Adolescents may participate in the 3-month interview if they did not participate in the 1-month interview. The team will select adolescents who report higher pain scores compared to peers undergoing similar procedures on the Weeks 1, 2 and 3 month surveys and a sample of adolescents who are recovering as anticipated. Interviews will take place via telephone or CHOP approved videoconferencing platform with transcription and transcripts, entered in REDCap, that only contain the patient's study identification (ID) as a personal identifier. It is anticipated that some adolescents will decline participation in the one-month survey; they will not be approached to participate in the three-month survey unless they indicate willingness to receive an invitation upon submitting the Month 3 survey. It is also anticipated that individuals may decline to participate in the three-month survey and Investigators will plan to extend additional invitations to complete approximately 25 interviews at each interval.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 11 to 21 years
2. Scheduled for non-cardiac surgery at one of five CHOP surgical centers
3. American Society of Anesthesiologists Physical Status (ASA) ≤ 3
4. Girls 11 years of age and older must have a negative urine/serum pregnancy test
5. Parental/guardian permission (informed consent) if participant <18 years old and if appropriate, child assent

Exclusion Criteria:

1. Subjects with limited English proficiency.
2. History of chronic pain
3. History of prior opioid use >5 consecutive days for acute pain or >10 consecutive days for major surgery in their life time
4. Pregnant or lactating females
5. Subjects who, in the opinion of the investigator, may be non-compliant with study schedules.

Ages: 11 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will enroll up to 500 adolescents age 11-21 years undergoing surgery at all CHOP surgical sites
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of new chronic pain | 7 months
  Incidence of new chronic pain, using the International Association for the Study of Pain (IASP) definition at 3 months after surgery, among a diverse cohort of adolescents undergoing major surgery. Prior reports in the adolescent surgery literature have suggested that 20% of patients develop chronic pain, defined as surgical site pain that persists more than three months after surgery. Here, Investigators have hypothesized that a lower chronic pain incidence of 11% exists among adolescents at CHOP after undergoing major surgery. Therefore using a two-sided Wald test to detect a significant difference from historic estimates, Investigators will enroll a minimum of 115 patients undergoing major surgery (a=0.05; b=0.1; n=95, assuming conservative 20% loss of follow-up). The remainder of the up to 500 subjects will represent a variety of procedures associated with mild, moderate and severe postoperative pain to characterize recovery trajectories.

SECONDARY OUTCOMES:
Prolonged opioid use compared to peers undergoing similar surgeries | 7 months
  Factors associated with prolonged opioid use after surgery, measured in time to opioid discontinuation after surgery, compared to peers undergoing similar surgeries
Delayed recovery compared to peers | 7 months
  Factors, including elevated average and maximum NRS scores, GAD-7 and PHQ-9 scores, and Screening to Brief Intervention (S2BI) scores, associated with delayed recovery from surgery compared to peers undergoing similar surgeries. For the NRS scale, which ranges from 0-10, a response of '0' corresponds to "no pain" while a response of '10' corresponds to extreme severe pain (e.g., "worst pain imaginable"). For the GAD-7 scale, a score of 5-9 corresponds to mild anxiety, 10-14 to moderate anxiety and 15+ to severe anxiety. For the PHQ-9 scale, 4 or more items selected in the shaded section corresponds to a possible depressive disorder with 5 or more corresponding to a possible major depressive disorder. For the S2BI scale, a never response corresponds to no reported substance use, once or twice corresponds to lower risk substance use and more than monthly corresponds to higher risk substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Tori N Sutherland, MD MPH, Principal Investigator — CHOP
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rabbitts JA, Palermo TM, Zhou C, Mangione-Smith R. Pain and Health-Related Quality of Life After Pediatric Inpatient Surgery. J Pain. 2015 Dec;16(12):1334-1341. doi: 10.1016/j.jpain.2015.09.005. Epub 2015 Sep 28. PMID 26416163
- [Background] Rabbitts JA, Fisher E, Rosenbloom BN, Palermo TM. Prevalence and Predictors of Chronic Postsurgical Pain in Children: A Systematic Review and Meta-Analysis. J Pain. 2017 Jun;18(6):605-614. doi: 10.1016/j.jpain.2017.03.007. Epub 2017 Mar 29. PMID 28363861
- [Background] Rabbitts JA, Palermo TM, Zhou C, Meyyappan A, Chen L. Psychosocial Predictors of Acute and Chronic Pain in Adolescents Undergoing Major Musculoskeletal Surgery. J Pain. 2020 Nov-Dec;21(11-12):1236-1246. doi: 10.1016/j.jpain.2020.02.004. Epub 2020 Jun 15. PMID 32553622
- [Background] Ward A, Jani T, De Souza E, Scheinker D, Bambos N, Anderson TA. Prediction of Prolonged Opioid Use After Surgery in Adolescents: Insights From Machine Learning. Anesth Analg. 2021 Aug 1;133(2):304-313. doi: 10.1213/ANE.0000000000005527. PMID 33939656
- [Background] Harbaugh CM, Lee JS, Chua KP, Kenney B, Iwashyna TJ, Englesbe MJ, Brummett CM, Bohnert AS, Waljee JF. Association Between Long-term Opioid Use in Family Members and Persistent Opioid Use After Surgery Among Adolescents and Young Adults. JAMA Surg. 2019 Apr 1;154(4):e185838. doi: 10.1001/jamasurg.2018.5838. Epub 2019 Apr 17. PMID 30810738
- [Background] Chua KP, Brummett CM, Conti RM, Bohnert A. Association of Opioid Prescribing Patterns With Prescription Opioid Overdose in Adolescents and Young Adults. JAMA Pediatr. 2020 Feb 1;174(2):141-148. doi: 10.1001/jamapediatrics.2019.4878. PMID 31841589
- [Background] Steinberg L. A Social Neuroscience Perspective on Adolescent Risk-Taking. Dev Rev. 2008 Mar;28(1):78-106. doi: 10.1016/j.dr.2007.08.002. PMID 18509515
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Rabbitts JA, Groenewald CB. Epidemiology of Pediatric Surgery in the United States. Paediatr Anaesth. 2020 Oct;30(10):1083-1090. doi: 10.1111/pan.13993. Epub 2020 Aug 29. PMID 32777147
- [Background] Harbaugh CM, Lee JS, Hu HM, McCabe SE, Voepel-Lewis T, Englesbe MJ, Brummett CM, Waljee JF. Persistent Opioid Use Among Pediatric Patients After Surgery. Pediatrics. 2018 Jan;141(1):e20172439. doi: 10.1542/peds.2017-2439. Epub 2017 Dec 4. PMID 29203521
- [Background] Rabbitts JA, Aaron RV, Fisher E, Lang EA, Bridgwater C, Tai GG, Palermo TM. Long-Term Pain and Recovery After Major Pediatric Surgery: A Qualitative Study With Teens, Parents, and Perioperative Care Providers. J Pain. 2017 Jul;18(7):778-786. doi: 10.1016/j.jpain.2017.02.423. Epub 2017 Feb 21. PMID 28232147
- [Background] Page MG, Stinson J, Campbell F, Isaac L, Katz J. Identification of pain-related psychological risk factors for the development and maintenance of pediatric chronic postsurgical pain. J Pain Res. 2013;6:167-80. doi: 10.2147/JPR.S40846. Epub 2013 Mar 5. PMID 23503375
- [Background] Sieberg CB, Simons LE, Edelstein MR, DeAngelis MR, Pielech M, Sethna N, Hresko MT. Pain prevalence and trajectories following pediatric spinal fusion surgery. J Pain. 2013 Dec;14(12):1694-702. doi: 10.1016/j.jpain.2013.09.005. PMID 24290449
- [Background] Page MG, Campbell F, Isaac L, Stinson J, Katz J. Parental risk factors for the development of pediatric acute and chronic postsurgical pain: a longitudinal study. J Pain Res. 2013 Sep 30;6:727-41. doi: 10.2147/JPR.S51055. eCollection 2013. PMID 24109194
- [Background] Rabbitts JA, Zhou C, Groenewald CB, Durkin L, Palermo TM. Trajectories of postsurgical pain in children: risk factors and impact of late pain recovery on long-term health outcomes after major surgery. Pain. 2015 Nov;156(11):2383-2389. doi: 10.1097/j.pain.0000000000000281. PMID 26381701
- [Background] Kharasch ED, Clark JD, Adams JM. Opioids and Public Health: The Prescription Opioid Ecosystem and Need for Improved Management. Anesthesiology. 2022 Jan 1;136(1):10-30. doi: 10.1097/ALN.0000000000004065. PMID 34874401
- [Background] Kelley-Quon LI, Kirkpatrick MG, Ricca RL, Baird R, Harbaugh CM, Brady A, Garrett P, Wills H, Argo J, Diefenbach KA, Henry MCW, Sola JE, Mahdi EM, Goldin AB, St Peter SD, Downard CD, Azarow KS, Shields T, Kim E. Guidelines for Opioid Prescribing in Children and Adolescents After Surgery: An Expert Panel Opinion. JAMA Surg. 2021 Jan 1;156(1):76-90. doi: 10.1001/jamasurg.2020.5045. PMID 33175130
- [Background] Chihuri S, Li G. Use of prescription opioids and motor vehicle crashes: A meta analysis. Accid Anal Prev. 2017 Dec;109:123-131. doi: 10.1016/j.aap.2017.10.004. Epub 2017 Oct 20. PMID 29059534
- [Background] Rabbitts JA, Kain Z. Perioperative Care for Adolescents Undergoing Major Surgery: A Biopsychosocial Conceptual Framework. Anesth Analg. 2019 Oct;129(4):1181-1184. doi: 10.1213/ANE.0000000000004048. No abstract available. PMID 30720491
- [Derived] Sutherland TN, Hadland SE, Moon J, Fardad J, Ramsay E, Kallan MJ, Neuman MD. The Adolescent Surgery Experience (ASE): a survey-based prospective cohort study to measure risk factors for persistent opioid use. BJA Open. 2025 Oct 15;16:100496. doi: 10.1016/j.bjao.2025.100496. eCollection 2025 Dec. PMID 41142590